CLINICAL TRIAL: NCT02175277
Title: Single Arm, Companion Study to Myelodysplastic Syndrome (MDS) 20090160 Using Darbepoetin Alfa for the Treatment of Anaemic Subjects With Myelodysplastic Syndrome
Brief Title: Darbepoetin Alfa MDS Companion Protocol
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20130113; 2013-000727-13 (EudraCT Number)
Record Dates: First submitted 2014-06-24; First posted 2014-06-26 (Estimated); Results first posted 2018-10-11 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-10

CONDITIONS: Myelodysplastic Syndrome (MDS)
Keywords: Myelodysplastic Syndrome (MDS); Darbepoetin alfa; low risk MDS; intermediate-1 risk MDS; International Prognostic Scoring System (IPSS)
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Darbepoetin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Darbepoetin Alfa (Experimental): Participants received darbepoetin alfa for up to 73 weeks or until progression to acute myeloid leukemia (AML), whichever occurred first.
  Interventions: Drug: Darbepoetin Alfa

INTERVENTIONS:
Drug: Darbepoetin Alfa — The first dose of darbepoetin alfa was the same as that administered at the last dosing visit of the active treatment period in Study 20090160. Doses could be increased up to a maximum of 500 μg every two weeks (Q2W).
  Other Names: Aranesp®

SUMMARY:
The primary objective of the study was to provide required access of investigational product (darbepoetin alfa) beyond the end of the active treatment period (EOATP) of the darbepoetin alfa MDS 20090160 (NCT01362140) study for patients who had continued demonstration of benefit from darbepoetin alfa treatment and to describe the safety of longer-term use in this patient population.

DETAILED DESCRIPTION:
This is a phase 3b, multi-centre, open-label, single-arm companion study to the MDS 20090160 study (NCT01362140) for the treatment of anaemic patients with MDS. Participants who completed the active-treatment period of the darbepoetin alfa MDS 20090160 study and met the eligibility criteria could be enrolled into this study to continue treatment of darbepoetin alfa for up to 73 weeks or until progression to acute myelogenous leukemia (AML), whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Subject or subject's legally acceptable representative has provided informed consent prior to any study-specific activities/ procedures being initiated;
* Subject must continue long term follow up within parent study (20090160);
* Subject must have an ongoing clinically relevant erythroid response as assessed by the Investigator using current response criteria (ie, International Working Group (IWG) response criteria);

Exclusion Criteria:

* Transfusion dependence defined as receiving a total of ≥ 4 units of red blood cell (RBC) transfusion in the previous 8-week period prior to enrolment;
* Known diagnosis of acute myelogenous leukemia (AML) or marrow collagen fibrosis;
* Known refractory anaemia with excess blast-2 (RAEB-2);
* Known diagnosis of intermediate-2 or high risk MDS per International Prognostic Scoring System (IPSS);
* Subjects received thrombopoiesis-stimulating factors (eg, eltrombopag, romiplostim) in the MDS 20090160 study or planning to receive such agents during the study;
* Other protocol defined inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-06-12 (Actual); Primary Completion 2017-03-20 (Actual); Study Completion 2017-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (4):
- Belgium (4):
  - Research Site, Charleroi
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Sint-Niklaas

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 5 centers in Belgium from 12 June 2014 (first participant enrolled) to 20 March 2017 (last participant completed study).
Pre-assignment Details: This study enrolled participants who completed the active treatment period of the phase 3 Study 20090160 (NCT01362140).
Period: Overall Study
Arm/Group | Darbepoetin Alfa
Started | 9
Completed | 8
Not Completed | 1
Not completed — Protocol-specified Criteria | 1

BASELINE CHARACTERISTICS:
Arm/Group | Darbepoetin Alfa
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.3 (7.9)
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 years | 1
  65 - 74 years | 6
  75 - 84 years | 2
  ≥ 85 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: Adverse events (AEs) were graded for severity according to the Common Terminology Criteria for Adverse Events (CTCAE), version 4.0, where Grade 1 indicates a mild AE, Grade 2 indicates a moderate AE, Grade 3 indicates severe or medically significant but not immediately life-threatening and Grade 4 indicates life-threatening consequences; urgent intervention indicated.
  A serious adverse event was defined as an adverse event that met at least one of the following serious criteria:
  * fatal
  * life threatening
  * required in-patient hospitalization or prolongation of existing hospitalization
  * resulted in persistent or significant disability/incapacity
  * congenital anomaly/birth defect
  * other medically important serious event The investigator assessed whether each adverse events was related to darbepoetin alfa.
Time Frame: From first dose of darbepoetin alfa to 30 days after last dose; the maximum treatment duration was 73 weeks.
Population: All enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Darbepoetin Alfa
Number analyzed (Participants) | 9
Participants
  All adverse events | 9
  Adverse events ≥ grade 2 | 8
  Adverse events ≥ grade 3 | 2
  Adverse events ≥ grade 4 | 0
  Serious adverse events | 3
  AEs leading to discontinuation of darbepoetin alfa | 1
  Fatal adverse events | 0
  Treatment-related adverse events | 0

ADVERSE EVENTS:
Time Frame: From first dose of darbepoetin alfa to 30 days after last dose; the maximum treatment duration was 73 weeks.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Darbepoetin Alfa
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 3/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Darbepoetin Alfa (N=9)
Macular fibrosis (Eye disorders) | 1
Pyrexia (General disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Darbepoetin Alfa (N=9)
Anaemia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
Chalazion (Eye disorders) | 1
Visual acuity reduced (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Aphthous ulcer (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Fatigue (General disorders) | 4
Injection site haematoma (General disorders) | 1
Malaise (General disorders) | 1
Pyrexia (General disorders) | 1
Bronchitis (Infections and infestations) | 1
Gingivitis (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 2
Oral fungal infection (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Restless legs syndrome (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1
Skin discomfort (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Haematoma (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Statistical Analysis Plan (2014-06-12): https://cdn.clinicaltrials.gov/large-docs/77/NCT02175277/SAP_001.pdf
  • Study Protocol (2013-04-15): https://cdn.clinicaltrials.gov/large-docs/77/NCT02175277/Prot_002.pdf